CLINICAL TRIAL: NCT01000493
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose Study Evaluating the Efficacy and Safety of the Neurokinin-1 Receptor Antagonist Orvepitant (GW823296) in Post Traumatic Stress Disorder (PTSD)
Brief Title: Orvepitant (GW823296) in Adult Post Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113211
Record Dates: First submitted 2009-10-15; First posted 2009-10-23 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-07

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: efficacy; double-blind; Clinician Administered PTSD Scale; placebo; Sleep; safety; CAPS; neurokinin-1 antagonist; orvepitant; PTSD; randomized; Post traumatic stress disorder; Phase II
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — orvepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orvepitant 60 mg (Experimental): 60 mg/day
  Interventions: Drug: orvepitant
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: orvepitant — Neurokinin-1 (NK-1) antagonist
  Other Names: GW823296
  Arms: Orvepitant 60 mg
Other: Placebo — Inactive placebo to match orvepitant 60 mg dosage form
  Arms: Placebo

SUMMARY:
This is a 12-week, randomized, multicenter, double-blind, placebo controlled, fixed-dose parallel group study to assess the efficacy and safety of orvepitant (60 mg/day) versus placebo in subjects with a diagnosis of noncombat-related Posttraumatic Stress Disorder (PTSD), whose symptoms are considered moderate or severe.

Following an initial screening visit, subjects fulfilling the study inclusion and exclusion criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and ECG assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. At the completion of the screening period, eligible subjects will be randomized at the baseline visit to receive either orvepitant 60mg/day or placebo (1:1 ratio). Those subjects randomized to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant.

Efficacy will be assessed using the Clinician Administered PTSD Scale (CAPS) as the primary efficacy measure. Key secondary efficacy endpoints will be based on the Davidson Trauma Scale (DTS), the Short PTSD Rating Interview (SPRINT), the Clinical Global Impression- Global Improvement and Severity of Illness Scales (CGI-I and CGI-S, respectively), the Hamilton Depression Rating Scale (HAM-D), the Cognitive and Physical Functioning Questionnaire (CPFQ) and the Pittsburgh Sleep Quality Index (PSQI).

Safety will be assessed by monitoring for adverse events (side effects) and through periodic laboratory evaluations (blood tests), vital signs assessments (e.g., blood pressure, heart rate, temperature) and heart function measurements (electrocardiograms, or ECGs).

DETAILED DESCRIPTION:
The purpose of the current study is to test the safety and effects of orvepitant, an investigational drug for the treatment of noncombat-related PTSD.

Efficacy will be assessed using standard symptom and severity rating scales (questionnaires). The Clinicain Adminstered PTSD Scale (CAPS) will serve as the primary measure of efficacy. Secondary efficacy endpoints include the CAPS subscale clusters (Re-Experiencing, Avoidance and Numbing, and Hyperarousal), the Davidson Trauma Scale (DTS), the Short PTSD Rating Interview (SPRINT), the Hamilton Depression Rating Scale (HAM-D), the Clinical Global Impression- Global Improvement and Severity of Illness Scale (CGI-I and CGI-S, respectively), the Cognitive and Physical Functioning Questionnaire (CPFQ) and the Pittsburgh Sleep Quality Index (PSQI).

Safety and tolerability will be assessed by monitoring adverse events (AEs or side effects), physical examinations (including vital signs such as blood pressure and heart rate), clinical laboratory assessments (blood tests), electrical recordings of the heart (electrocardiograms or ECG's), the Columbia Suicidality Severity Rating Scale (CSSRS), Massachusetts Sexual Function Questionnaire (MSFQ), Discontinuation-Emergent Signs and Symptoms (DESS) scale and weight change.

Blood samples will be taken at different time points to assess blood levels of orvepitant in patients, allowing the relationship between amount of orvepitant in the body and efficacy to be studied.

The primary objective of the study is to evaluate the efficacy of orvepitant (60mg/day) versus placebo (a "sugar pill", with no active ingredients). The secondary objectives include assessing the safety and tolerability of orvepitant, assessing the profile of appearance and disappearance of orvepitant in the body (blood) following administration (i.e., assessing how long the drug remains in the body), and lastly to examine the relationship between blood levels of the drug and efficacy (i..e, the change in CAPS score relative to what it was before starting the study medication).

Following an initial screening visit, subjects fulfilling the study entrance criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and electrocardiogram assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. Upon completion of the screening period, eligible subjects will be randomly assigned at the baseline visit to one of two treatment regimens: orvepitant 60mg/day or placebo for a 12-week treatment phase. The chances of receiving each of the two possible treatments will be equal. Orvepitant will be administered as tablets. Those subjects randomised to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant.

During the treatment phase, subjects will be required to return to the clinic at the end of Weeks 1, 2, 4, 6, 8, 10 and 12. In addition, all subjects will be required to return for a follow-up visit 14 days after the last dose of study medication. In addition, all subjects with ongoing adverse events at the 14-day follow-up visit will be required to return for a further follow-up visit 28 days after the last dose of study medication. Women of child-bearing potential will also be required to attend the 28-Day follow-up visit for a pregnancy test. A further test will be performed 42 Days following the end of treatment.

Male and female outpatients between the ages of 18 to 64 years inclusive with a primary diagnosis of noncombat-related PTSD will be enrolled into this study. A total of approximately 240 subjects are expected to be enrolled at approximately 25 different study sites in North America.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years, inclusive.
* A primary diagnosis of noncombat-related Post traumatic Stress Disorder (PTSD)
* Subjects with symptom severity considered to be at least moderate to severe.

Exclusion Criteria:

* Subjects whose symptoms are better accounted for by a diagnosis other than Post traumatic Stress Disorder (PTSD), subjects diagnosed with dementia; subjects diagnosed with a current/recent eating disorder such as anorexia nervosa or bulimia; subjects with a diagnosed history of schizophrenia, schizoaffective disorder, or Bipolar Disorder.
* Subjects who have a history of failing to respond to adequate treatment for PTSD with an antidepressant/anti-anxiety drug, i..e, failure to improve following administration of at least two other antidepressants/anti-anxiety drugs, each given for at least 4 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2009-11-02 (Actual); Primary Completion 2010-06-28 (Actual); Study Completion 2010-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (26):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Weymouth, Massachusetts
  - GSK Investigational Site, Willingboro, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Garfield Heights, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Brown Deer, Wisconsin
  - GSK Investigational Site, Middleton, Wisconsin

REFERENCES:
- [Background] Ratti E, Bettica P, Alexander R, Archer G, Carpenter D, Evoniuk G, Gomeni R, Lawson E, Lopez M, Millns H, Rabiner EA, Trist D, Trower M, Zamuner S, Krishnan R, Fava M. Full central neurokinin-1 receptor blockade is required for efficacy in depression: evidence from orvepitant clinical studies. J Psychopharmacol. 2013 May;27(5):424-34. doi: 10.1177/0269881113480990. Epub 2013 Mar 28. PMID 23539641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 participants with posttraumatic stress disorder were randomized to either orvepitant (GW823296) 60 milligrams (mg) or placebo at 26 centres in the United States. Intention to treat (ITT) population included total of 120 participants.
Pre-assignment Details: The study was prematurely terminated on 11 May 2010 upon the recommendation of the Data Safety Monitoring Board.
Groups:
- Placebo: Participants assigned to take one tablet of matching placebo of orvepitant each day in the evening (once daily) up to 12 weeks.
- Orvepitant 60 mg Once Daily: Participants assigned to take one tablet of orvepitant 60 mg each day in the evening (once daily) up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Started | 60 | 69
Completed | 21 | 14
Not Completed | 39 | 55
Not completed — Adverse Event | 3 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 1 | 8
Not completed — Study closed/terminated | 25 | 23
Not completed — Lost to Follow-up | 5 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Orvepitant 60 mg Once Daily | Total
Number analyzed (Participants) | 60 | 69 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (10.88) | 37.0 (12.24) | 36.7 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 13 | 17 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 20 | 37
  White | 38 | 48 | 86
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 17-item Clinician Administered Posttraumatic Stress Disorder (PTSD) Scale (CAPS) Total Severity Score at Week 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS total severity score was based on the 17 items that assess the frequency and intensity of PTSD symptoms. There were 8 items assessing associated features (guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment). The total score 0-136, higher scores means more severity, < 20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and > 80: extreme PTSD symptoms. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and Week 12
Population: ITT population, consisted of all participants who gave informed consent, were randomized, received at least one dose of double blind medication and for whom at least one post-randomization assessment was available. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 21 | 14
Score on scale | -25.75 (4.084) | -31.38 (4.611)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3624, MMRM analysis — The mixed effects model repeated measures (MMRM) analysis included treatment, week, Baseline total CAPS score and the treatment by week and Baseline. Week was used as the repeated effect in the model; Mean Difference (Net) = -5.62, 95% CI 2-sided [-17.9 to 6.65] — Comparison between Placebo and Orvepitant 60 mg at Week 12

2. Secondary Outcome: Percentage of Participants Responding, Based on More Than Equal to (>=) 30 Percent (%) Reduction From Baseline in CAPS Total Severity Score at Weeks 1, 4, 8 and 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS total severity score was based on the 17 items that assess the frequency and intensity of PTSD symptoms. There were 8 items assessing associated features (guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment). The total score 0-136, higher scores means more severity, < 20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and > 80: extreme PTSD symptoms. Percentage of participants were calculated by total number of responders divided by number of participants assessed multiplied by 100.
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | 7 | 13
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | 50 | 38
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | 47 | 68
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | 52 | 79
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3156, Logistic regression analysis; The analysis method was logistic regression adjusted for Baseline CAPS total score; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.54 to 6.76] — Comparison between Placebo and Orvepitant 60 mg at Week 1. Odds ratios represent the odds of improvement, relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3024, Logistic regression analysis; The analysis method was logistic regression adjusted for Baseline CAPS total score; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.27 to 1.50] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1208, Logistic regression analysis; The analysis method was logistic regression adjusted for Baseline CAPS total score; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.79 to 7.28] — Comparison between Placebo and Orvepitant 60 mg at Week 8. Odds ratios represent the odds of improvement, relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1331, Logistic regression analysis; The analysis method was logistic regression adjusted for Baseline CAPS total score; Odds Ratio (OR) = 3.27, 95% CI 2-sided [0.70 to 15.4] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: The Time to (Maintained) Clinical Response in Each Participants
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS total severity score was based on the 17 items that assess the frequency and intensity of PTSD symptoms. There were 8 items assessing associated features (guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment). The total score 0-136, higher scores means more severity, < 20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and > 80: extreme PTSD symptoms. The time required to maintain CAPS response has been summarized.
Time Frame: Up to Week 12
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 10 | 9
Days | 35.5 [29.0 to 58.0] | 30.0 [28.0 to 57.0]

4. Secondary Outcome: Change From Baseline in the 17-item CAPS Total Severity Score at Weeks 1, 4, and 8
Description: as for outcome 1
Time Frame: Baseline (Day 1 pre-dose) and Week 1, 4, 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -9.24 (1.640) | -10.11 (1.562)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -24.24 (2.566) | -21.43 (2.430)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -23.33 (3.572) | -27.97 (3.704)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.7015, MMRM analysis — The MMRM analysis model included treatment, week, Baseline total CAPS score, and the treatment by week and Baseline by week interaction terms. Week was used as the repeated effect in the model; Mean Difference (Net) = -0.87, 95% CI 2-sided [-5.35 to 3.61] — Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.4292, MMRM analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = 2.81, 95% CI 2-sided [-4.22 to 9.84] — Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3702, MMRM analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -4.64, 95% CI 2-sided [-14.9 to 5.62] — Comparison between placebo and orvepitant 60 mg once daily at Week 8

5. Secondary Outcome: Percentage of Participants Remitting, Based on a CAPS Total Score < 20 at Weeks 1, 4, 8, and 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS total severity score was based on the 17 items that assess the frequency and intensity of PTSD symptoms. There were 8 items assessing associated features (guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment). The total score 0-136, higher scores means more severity, < 20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and > 80: extreme PTSD symptoms. Remitter defined as a participants who has a CAPS total score <20. Percentage of participants were calculated by total number of responders divided by number of participants assessed multiplied by 100.
Time Frame: Up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed. The analysis method was logistic regression adjusted for Baseline CAPS total score. At a visit where there were no remitters, no analysis was performed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | 0 | 0
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | 5 | 2
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | 3 | 4
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | 10 | 7
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.5719, Logistic regression analysis; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.04 to 5.82] — Odds ratios represent the odds of improvement, relative to place. Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9080, Logistic regression analysis; Odds Ratio (OR) = 1.18, 95% CI [0.07 to 20.1] — Odds ratios represent the odds of improvement, relative to place. Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9486, Logistic regression analysis; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.07 to 12.5] — Odds ratios represent the odds of improvement, relative to place. Comparison between placebo and orvepitant 60 mg once daily at Week 12

6. Secondary Outcome: Change From Baseline in the CAPS Re-experiencing Subscale Cluster Score at Weeks 1, 4, 8 and 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS assessed Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnostic criteria for PTSD, including criteria B-D (core symptom clusters of re-experiencing). The re-experiencing subscale cluster score was derived from the CAPS. The possible range was 5 to 25 with lower score indicates less severe symptoms and with a greater score indicating greater PTSD symptom severity. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -3.1 (5.91) | -4.6 (5.96)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -8.4 (7.77) | -8.0 (6.50)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -8.5 (8.50) | -10.0 (7.85)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -10.0 (8.75) | -12.9 (10.50)

7. Secondary Outcome: Change From Baseline in the CAPS Avoidance/Numbing (A/N) Subscale Cluster Score at Weeks 1, 4, 8, and 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS assessed DSM-IV diagnostic criteria for PTSD, including criteria B-D (core symptom clusters of A/N). The re-experiencing subscale cluster score was derived from the CAPS. The possible range is 7 to 35 with lower score indicates less severe symptoms and with a greater score indicating greater PTSD symptom severity. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -3.22 (0.791) | -2.55 (0.757)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -8.99 (1.180) | -8.48 (1.122)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -7.74 (1.734) | -9.96 (1.817)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -9.13 (1.906) | -11.11 (2.143)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.5426, MMRM analysis — The MMRM analysis model included treatment, week, Baseline CAPS A/N subscore and the treatment by week and Baseline by week interaction terms. Week was used as the repeated effect in the model; Mean Difference (Net) = 0.67, 95% CI 2-sided [-1.51 to 2.85] — Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.7552, MMRM analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.51, 95% CI 2-sided [-2.73 to 3.75] — Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3827, MMRM analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -2.22, 95% CI 2-sided [-7.27 to 2.83] — Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.4915, MMRM analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -1.98, 95% CI 2-sided [-7.71 to 3.75] — Comparison between placebo and orvepitant 60 mg once daily at Week 12

8. Secondary Outcome: Change From Baseline in the CAPS Hyperarousal Subscale Cluster Score at Weeks 1, 4, 8, and 12
Description: The CAPS was a 30-item clinical interview. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The CAPS assessed DSM-IV diagnostic criteria for PTSD, including criteria B-D (core symptom clusters of hyperarousal). The re-experiencing subscale cluster score was derived from the CAPS. The possible range is 5 to 25 with lower score indicates less severe symptoms and with a greater score indicating greater PTSD symptom severity. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -2.86 (0.672) | -2.96 (0.639)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -6.66 (0.982) | -5.34 (0.930)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -7.26 (1.324) | -7.33 (1.394)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -8.02 (1.388) | -8.93 (1.689)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9190, MMRM analysis — The MMRM analysis model included treatment, week, Baseline CAPS hyperarousal subscore and the treatment by week and Baseline by week interaction terms. Week was used as the repeated effect in the model; Mean Difference (Net) = -0.09, 95% CI 2-sided [-1.93 to 1.74] — Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.3326, MMRM analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-1.37 to 4.00] — Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9712, MMRM analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-3.91 to 3.77] — Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.6711, MMRM analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Net) = -0.92, 95% CI 2-sided [-5.22 to 3.39] — Comparison between placebo and orvepitant 60 mg once daily at Week 12

9. Secondary Outcome: Percentage of Participants Responding, Based on a Clinical Global Impression- Global Improvement (CGI-I) Score of 1 or 2, by Visit Week
Description: The global improvement items were rated on a 1-7 scale with 0 means not assessed (1: very much improved, 2: much improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: much worse, 7: very much worse). For the global improvement item, the clinician indicated their assessment of the participant's total improvement or worsening compared with that individual's condition at the start of the study (the Baseline visit) whether or not the change was judged to be due to drug treatment. Responder was defined as a participant who had a CGI-I score of 1 or 2 ('very much improved' or 'much improved'). It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. Percentage of participants were calculated by total number of responders divided by number of participants assessed multiplied by 100.
Time Frame: Up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Percentage of participants
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | 5 | 8
  Week 2: number analyzed (Participants) | 53 | 58
  Week 2 | 15 | 21
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | 29 | 30
  Week 6: number analyzed (Participants) | 37 | 33
  Week 6 | 35 | 58
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | 33 | 48
  Week 10: number analyzed (Participants) | 27 | 21
  Week 10 | 30 | 57
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | 43 | 71
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.5532, Logistic regression analysis — The analysis method was logistic regression adjusted for Baseline total Clinical Global Impression-Severity of Illness scales (CGI-S) score; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.36 to 6.92] — Odds ratios represent the odds of improvement, relative to placebo. Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.4508, Logistic regression analysis; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.54 to 3.93] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 2
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9234, Logistic regression analysis; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.42 to 2.62] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0662, Logistic regression analysis; Odds Ratio (OR) = 2.48, 95% CI 2-sided [0.94 to 6.53] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.2767, Logistic regression analysis; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.61 to 5.48] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0588, Logistic regression analysis; Odds Ratio (OR) = 3.17, 95% CI 2-sided [0.96 to 10.5] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 10
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1032, Logistic regression analysis; Odds Ratio (OR) = 3.33, 95% CI 2-sided [0.78 to 14.1] — Odds ratios represent the odds of improvement, relative to placebo. The analysis method was logistic regression adjusted for Baseline total CGI-S score. Comparison between placebo and orvepitant 60 mg once daily at Week 12

10. Secondary Outcome: Change From Baseline in the CGI-S Score, by Visit Week
Description: The severity of illness items were rated on a 1-7 scale with 0 means not assessed (1: normal, not at all ill, 2: borderline mentally ill, 3: mildly ill, 4: moderately ill, 5: markedly ill, 6: severely ill, 7: among the most extremely ill participants). For the severity of illness item, the clinician indicated his/her assessment of the participant severity of illness considering their total clinical experience with the particular population being studied. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -0.23 (0.064) | -0.35 (0.061)
  Week 2: number analyzed (Participants) | 53 | 58
  Week 2 | -0.44 (0.093) | -0.65 (0.089)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -0.84 (0.127) | -0.84 (0.120)
  Week 6: number analyzed (Participants) | 37 | 33
  Week 6 | -0.73 (0.140) | -1.03 (0.140)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -0.67 (0.150) | -1.28 (0.155)
  Week 10: number analyzed (Participants) | 27 | 21
  Week 10 | -0.83 (0.188) | -1.26 (0.195)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -1.10 (0.195) | -1.42 (0.216)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1743, MMRM analysis — The MMRM analysis model included treatment, week, baseline CGI-S score, and the treatment by week and baseline by week interaction terms. Week was used as the repeated effect in the model; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.29 to 0.05] — Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1181, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.46 to 0.05] — Comparison between placebo and orvepitant 60 mg once daily at Week 2
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.9698, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.35 to 0.34] — Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1341, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.69 to 0.09] — Comparison between placebo and orvepitant 60 mg once daily at Week 6
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0064, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.04 to -0.18] — Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1095, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.98 to 0.10] — Comparison between placebo and orvepitant 60 mg once daily at Week 10
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.2814, MMRM analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.90 to 0.27] — Comparison between placebo and orvepitant 60 mg once daily at Week 12

11. Secondary Outcome: Change From Baseline in the Short PTSD Rating Review (SPRINT), by Visit Week
Description: The SPRINT consists of 8 items that assess the core symptoms of PTSD, as well as related aspects of somatic malaise, stress vulnerability and functional impairment. Each item was rated on a 5 point scale (0: not at all, 1: a little bit, 2: moderately, 3: quiet a lot and 4: very much), total score 0-32; with higher scores means more severity. Also, it provided the information about how the participant feeling (as a percentage) and symptoms improved since beginning of treatment (rated on a 5 point scale [0: worse, 1: a no change, 2: minimally, 3: much and 4: very much]). The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -2.1 (4.30) | -2.1 (4.69)
  Week 2: number analyzed (Participants) | 53 | 58
  Week 2 | -3.1 (5.44) | -5.1 (5.63)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -4.5 (6.24) | -4.9 (6.68)
  Week 6: number analyzed (Participants) | 37 | 33
  Week 6 | -4.6 (5.85) | -7.5 (7.24)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -6.0 (5.89) | -8.2 (6.56)
  Week 10: number analyzed (Participants) | 27 | 21
  Week 10 | -6.0 (6.80) | -8.1 (7.34)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -7.8 (6.66) | -8.8 (7.23)

12. Secondary Outcome: Change From Baseline in the Self-rated Davidson Trauma Scale (DTS), by Visit Week
Description: This instrument consists of 17 items which parallel the DSM criteria for PTSD. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) rated using 5-point scale. There were 8 items assessing associated features (guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment). The DTS cluster includes intrusion (items 1-4, 17 [score 0-40]), avoidance/numbing (A/N; items 5-11 [score 0-56]) and hyperarousal (items 12-16 [score 0-40]). The total score (0-136) was added, lower score indicates less symptoms and higher scores means more severity, <20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and > 80: extreme PTSD symptoms. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 55 | 61
  Week 1 | -11.3 (19.00) | -17.7 (20.60)
  Week 2: number analyzed (Participants) | 52 | 57
  Week 2 | -18.3 (22.64) | -25.4 (24.00)
  Week 4: number analyzed (Participants) | 41 | 46
  Week 4 | -24.7 (27.76) | -26.5 (24.36)
  Week 6: number analyzed (Participants) | 36 | 32
  Week 6 | -21.3 (29.04) | -36.1 (22.27)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -27.8 (27.58) | -42.9 (24.41)
  Week 10: number analyzed (Participants) | 27 | 21
  Week 10 | -25.3 (26.46) | -40.4 (32.88)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -33.3 (29.97) | -51.9 (25.73)

13. Secondary Outcome: Change From Baseline in the DTS Cluster Sub Score
Description: This instrument consists of 17 items which parallel the DSM criteria for PTSD. Both frequency (0: never; 4: daily or all the time) and intensity (0: none or no problem; 4: extreme, incapacitating) rated using 5-point scale and added to get total score. There were 8 items including guilt, hopelessness, memory impairment, overall response validity, global PTSD severity, global improvement and social and occupational impairment. The DTS cluster includes intrusion (items 1-4, 17 [score 0-40]), A/N (items 5-11 [score 0-56]) and hyperarousal (items 12-16 [score 0-40]) with lower score indicates less symptoms and higher scores means more severity, <20: few symptoms or being asymptomatic, 20-39: mild or subthreshold PTSD, 40-59: threshold and moderate PTSD, 60-79: severe PTSD symptoms and >80: extreme PTSD symptoms. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Intrusion, Week 1: number analyzed (Participants) | 55 | 61
  Intrusion, Week 1 | -4.7 (7.98) | -5.8 (7.56)
  Intrusion, Week 2: number analyzed (Participants) | 52 | 57
  Intrusion, Week 2 | -5.6 (8.10) | -7.9 (7.57)
  Intrusion, Week 4: number analyzed (Participants) | 41 | 46
  Intrusion, Week 4 | -8.4 (9.33) | -8.7 (8.25)
  Intrusion, Week 6: number analyzed (Participants) | 36 | 32
  Intrusion, Week 6 | -6.1 (8.76) | -10.0 (7.92)
  Intrusion, Week 8: number analyzed (Participants) | 30 | 25
  Intrusion, Week 8 | -8.3 (8.84) | -12.5 (8.62)
  Intrusion, Week 10: number analyzed (Participants) | 27 | 21
  Intrusion, Week 10 | -7.0 (7.75) | -12.5 (12.02)
  Intrusion, Week 12: number analyzed (Participants) | 21 | 14
  Intrusion, Week 12 | -10.0 (8.23) | -15.7 (10.93)
  A/N, Week 1: number analyzed (Participants) | 55 | 61
  A/N, Week 1 | -2.8 (8.91) | -5.2 (10.00)
  A/N, Week 2: number analyzed (Participants) | 52 | 57
  A/N, Week 2 | -6.7 (10.91) | -8.7 (11.76)
  A/N, Week 4: number analyzed (Participants) | 41 | 46
  A/N, Week 4 | -8.6 (15.06) | -9.1 (11.82)
  A/N, Week 6: number analyzed (Participants) | 36 | 32
  A/N, Week 6 | -7.8 (15.62) | -13.0 (10.96)
  A/N, Week 8: number analyzed (Participants) | 30 | 25
  A/N, Week 8 | -11.0 (13.22) | -16.2 (11.87)
  A/N, Week 10: number analyzed (Participants) | 27 | 21
  A/N, Week 10 | -10.1 (12.77) | -14.6 (13.88)
  A/N, Week 12: number analyzed (Participants) | 21 | 14
  A/N, Week 12 | -13.2 (15.59) | -19.9 (9.89)
  Hyperarousal, Week 1: number analyzed (Participants) | 55 | 61
  Hyperarousal, Week 1 | -3.8 (7.39) | -6.8 (7.41)
  Hyperarousal, Week 2: number analyzed (Participants) | 52 | 57
  Hyperarousal, Week 2 | -5.9 (8.41) | -8.7 (8.09)
  Hyperarousal, Week 4: number analyzed (Participants) | 41 | 46
  Hyperarousal, Week 4 | -7.6 (8.49) | -8.7 (8.67)
  Hyperarousal, Week 6: number analyzed (Participants) | 36 | 32
  Hyperarousal, Week 6 | -7.4 (8.08) | -13.0 (8.11)
  Hyperarousal, Week 8: number analyzed (Participants) | 30 | 25
  Hyperarousal, Week 8 | -8.5 (9.67) | -14.2 (7.54)
  Hyperarousal, Week 10: number analyzed (Participants) | 27 | 21
  Hyperarousal, Week 10 | -8.2 (9.41) | -13.3 (9.93)
  Hyperarousal, Week 12: number analyzed (Participants) | 21 | 14
  Hyperarousal, Week 12 | -10.1 (9.31) | -16.3 (9.46)

14. Secondary Outcome: Change From Baseline in the Pittsburgh Sleep Quality Index (PSQI) Global Score, by Visit Week
Description: The PSQI was a self-rated questionnaire to assess sleep quality and disturbances. Individual items (19) generate 7-component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. The global score generated by addition of individual score excluding use of sleeping medication component. It contains 15 objective (about frequency of sleep disturbances and subjective sleep quality) and 4 subjective (typical bedtime, wake-up time, sleep latency and sleep duration) items with score range from 0: no to 3: severe difficulty. The PSQI Global Score ranges from 0 to 21 and a global score > 5 was suggestive of significant sleep disturbance. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 53 | 58
  Week 1 | -1.6 (3.81) | -3.2 (4.11)
  Week 2: number analyzed (Participants) | 50 | 56
  Week 2 | -2.0 (3.71) | -4.3 (4.50)
  Week 4: number analyzed (Participants) | 37 | 42
  Week 4 | -3.2 (4.60) | -3.5 (4.72)
  Week 6: number analyzed (Participants) | 34 | 32
  Week 6 | -3.5 (4.02) | -4.3 (4.71)
  Week 8: number analyzed (Participants) | 27 | 23
  Week 8 | -3.2 (4.57) | -5.2 (4.69)
  Week 10: number analyzed (Participants) | 26 | 20
  Week 10 | -3.5 (5.11) | -4.6 (4.35)
  Week 12: number analyzed (Participants) | 20 | 14
  Week 12 | -4.6 (5.34) | -4.1 (5.21)

15. Secondary Outcome: Change From Baseline in the PSQI Addendum for PTSD (PSQI-A) Global Score, by Visit Week
Description: The PSQI-A was self-report instrument to assess disruptive nocturnal behavior (DNB) in PTSD participants with 7 types of DNB. These items include frequency of 1: hot flashes, 2: general nervousness, 3: memories or nightmares of traumatic experience, 4: severe anxiety or panic, not related to traumatic memories, 5: bad dreams, not related to traumatic memories, 6: episodes of terror or screaming during sleep without fully awakening and 7: episodes of acting out dreams, such as kicking, punching, running, or screaming. Each item was rated on a scale (0: not in the past month, 1: less than once a week, 2: once or twice a week and 3: three or more times a week) with global score range of 0-21. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 1 | 0
  Week 1 | -1.0 (NA) — SD was not derived as one participant was present at this time point. |
  Week 2: number analyzed (Participants) | 5 | 2
  Week 2 | -2.6 (2.07) | 0.5 (7.78)
  Week 4: number analyzed (Participants) | 41 | 46
  Week 4 | -1.9 (3.57) | -2.8 (3.58)
  Week 6: number analyzed (Participants) | 5 | 5
  Week 6 | 0.0 (2.55) | -7.0 (6.75)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -2.2 (3.99) | -4.0 (4.85)
  Week 10: number analyzed (Participants) | 4 | 6
  Week 10 | 1.5 (3.32) | -1.7 (6.35)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -3.3 (4.27) | -3.6 (4.83)

16. Secondary Outcome: Change From Baseline in the CAPS Recurrent Distressing Dreams Item (B2) at Weeks 1, 4, 8, and 12
Description: The B2 asked participant about 'Have you ever had unpleasant dreams about the event(s)? How often in the past month?' Both frequency (0: never; 4: daily or all the time) and 'at their worst, how much distress or discomfort did these dreams cause you? Did these dreams wake you up? [If yes, ask:] What were you feeling or doing when you awoke? How long does it usually take to get back to sleep? [Listen for report of panic symptoms, yelling, posturing] intensity (0: none or no problem with symptoms; 4: extreme, incapacitating) ratings were made on a 5-point scale. The total score 0-8, higher scores means more severity. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -1.2 (2.47) | -1.0 (2.48)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -1.4 (2.72) | -1.7 (2.48)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -1.9 (2.65) | -2.3 (3.12)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -1.4 (3.25) | -2.4 (3.10)

17. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HAM-D), by Visit Week
Description: The HAM-D was observer-rated depressive symptom rating scale to measure the severity of depressive symptoms in participants with primary depressive illness. The items were ranked on a scale of 0-4 (0: absent; 4: greatest severity) or 0-2 (0: no difficulty; 2: difficulty falling asleep). In addition to the total score (0-66; with higher score indicates more depression), the HAM-D anxiety factor score (sum of items 10, 11, 12, 13, 15 and 17) and the melancholia subscore (sum of items 1, 2, 7, 8, 10, and 13) of the 17-item HAM-D scale was analyzed. The melancholia subscale was derived from three formal psychometric criteria (calibration, ascending monotonicity and dispersion). It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 56 | 62
  Week 1 | -1.72 (0.518) | -3.64 (0.491)
  Week 2: number analyzed (Participants) | 53 | 58
  Week 2 | -3.42 (0.645) | -5.36 (0.613)
  Week 4: number analyzed (Participants) | 42 | 47
  Week 4 | -3.57 (0.866) | -5.46 (0.819)
  Week 6: number analyzed (Participants) | 37 | 33
  Week 6 | -3.73 (0.865) | -6.62 (0.865)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -3.83 (1.030) | -6.69 (1.061)
  Week 10: number analyzed (Participants) | 27 | 21
  Week 10 | -4.53 (1.143) | -7.41 (1.215)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -6.21 (1.341) | -6.48 (1.507)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0083, MMRM analysis — The MMRM analysis model included treatment, week, Baseline total HAM-D score, and the treatment by week and Baseline by week interaction terms. Week was used as the repeated effect in the model; Mean Difference (Net) = -1.92, 95% CI 2-sided [-3.33 to -0.50] — Comparison between placebo and orvepitant 60 mg once daily at Week 1
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0311, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.94, 95% CI 2-sided [-3.71 to -0.18] — Comparison between placebo and orvepitant 60 mg once daily at Week 2
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.1155, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -1.89, 95% CI 2-sided [-4.26 to 0.47] — Comparison between placebo and orvepitant 60 mg once daily at Week 4
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0210, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -2.89, 95% CI 2-sided [-5.33 to -0.45] — Comparison between placebo and orvepitant 60 mg once daily at Week 6
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0582, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -2.86, 95% CI 2-sided [-5.83 to 0.10] — Comparison between placebo and orvepitant 60 mg once daily at Week 8
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.0927, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -2.88, 95% CI 2-sided [-6.25 to 0.49] — Comparison between placebo and orvepitant 60 mg once daily at Week 10
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 60 mg Once Daily; Test type: Superiority or Other; p = 0.8954, MMRM analysis — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Net) = -0.27, 95% CI 2-sided [-4.36 to 3.83] — Comparison between placebo and orvepitant 60 mg once daily at Week 12

18. Secondary Outcome: Change From Baseline in the Cognitive and Physical Function Questionnaire (CPFQ) Total Score, by Visit Week
Description: The Massachusetts CPFQ was a brief self-report scale to measure cognitive and executive dysfunction in mood and anxiety disorders. The CPFQ comprises 7 questions assessing each of the most common complaints of depressed participants reporting fatigue or cognitive/executive problems. Each question was rated on a scale of 1 to 6, with 1: greater than normal, 2: normal, 3: minimally diminished, 4: moderately diminished, 5: markedly diminished and 6: totally absent functioning with total score 7-42; higher score indicating more dysfunction. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 56 | 64
Score on a scale
  Week 1: number analyzed (Participants) | 1 | 0
  Week 1 | 5.0 (NA) — SD was not derived as one participant was present at this time point. |
  Week 2: number analyzed (Participants) | 5 | 2
  Week 2 | -1.6 (4.72) | -2.5 (2.12)
  Week 4: number analyzed (Participants) | 41 | 46
  Week 4 | -2.0 (4.77) | -2.2 (7.29)
  Week 6: number analyzed (Participants) | 5 | 5
  Week 6 | -0.8 (5.26) | -5.2 (6.30)
  Week 8: number analyzed (Participants) | 30 | 25
  Week 8 | -3.9 (5.11) | -4.0 (7.38)
  Week 10: number analyzed (Participants) | 4 | 6
  Week 10 | 1.0 (4.55) | -0.8 (14.33)
  Week 12: number analyzed (Participants) | 21 | 14
  Week 12 | -5.3 (5.52) | -4.2 (6.76)

19. Secondary Outcome: Change From Baseline in Massachusetts Sexual Function Questionnaire (MSFQ) Total Score and Erectile Dysfunction Score in Males
Description: The MSFQ was derived from the Guided Interview Questionnaire for males and from the Arizona Sexual Experience Scale. The questionnaire includes five items with a score ranging from 1-6 (1: greater than normal; 2: normal; 3: minimally diminished; 4: moderately diminished; 5: markedly diminished and 6: totally absent with total score 5-30; higher score indicating more dysfunction). The areas of sexual functioning included were total score and erectile dysfunction (males only). A total score was used as a global measure of sexual dysfunction. A follow-up version of the questionnaire includes an additional sixth item of the participant's global impression of improvement, with a score ranging from 1 to 6. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: Male participants from all subject population used. All subject population defined as participants who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 13 | 17
Score on a scale
  Total score, Week 1: number analyzed (Participants) | 1 | 0
  Total score, Week 1 | -1.0 (NA) — SD was not derived as one participant was present at this time point. |
  Total score, Week 2: number analyzed (Participants) | 3 | 0
  Total score, Week 2 | -2.3 (6.03) |
  Total score, Week 4: number analyzed (Participants) | 8 | 11
  Total score, Week 4 | 0.1 (2.03) | -0.6 (5.48)
  Total score, Week 6: number analyzed (Participants) | 1 | 3
  Total score, Week 6 | 7.0 (NA) — SD was not derived as one participant was present at this time point. | 1.0 (1.73)
  Total score, Week 8: number analyzed (Participants) | 5 | 9
  Total score, Week 8 | -1.2 (2.77) | -3.7 (5.59)
  Total score, Week 10: number analyzed (Participants) | 1 | 3
  Total score, Week 10 | -1.0 (NA) — SD was not derived as one participant was present at this time point. | -7.3 (6.11)
  Total score, Week 12: number analyzed (Participants) | 3 | 6
  Total score, Week 12 | 2.0 (9.17) | -3.2 (6.62)
  Erectile dysfunction score, Week 1: number analyzed (Participants) | 1 | 0
  Erectile dysfunction score, Week 1 | 0.0 (NA) — SD was not derived as one participant was present at this time point. |
  Erectile dysfunction score, Week 2: number analyzed (Participants) | 3 | 0
  Erectile dysfunction score, Week 2 | -0.3 (0.58) |
  Erectile dysfunction score, Week 4: number analyzed (Participants) | 8 | 11
  Erectile dysfunction score, Week 4 | 0.1 (0.64) | -0.3 (1.56)
  Erectile dysfunction score, Week 6: number analyzed (Participants) | 1 | 3
  Erectile dysfunction score, Week 6 | 1.0 (NA) — SD was not derived as one participant was present at this time point. | -0.3 (0.58)
  Erectile dysfunction score, Week 8: number analyzed (Participants) | 5 | 9
  Erectile dysfunction score, Week 8 | -0.2 (0.45) | -0.7 (1.12)
  Erectile dysfunction score, Week 10: number analyzed (Participants) | 1 | 3
  Erectile dysfunction score, Week 10 | -1.0 (NA) — SD was not derived as one participant was present at this time point. | -1.3 (1.53)
  Erectile dysfunction score, Week 12: number analyzed (Participants) | 3 | 6
  Erectile dysfunction score, Week 12 | 0.3 (1.53) | -0.8 (1.33)

20. Secondary Outcome: Change From Baseline in MSFQ Total Score in Females
Description: The MSFQ was derived from the Guided Interview Questionnaire for males and from the Arizona Sexual Experience Scale. The questionnaire includes five items with a score ranging from 1-6 (1: greater than normal; 2: normal; 3: minimally diminished; 4: moderately diminished; 5: markedly diminished and 6: totally absent with total score 5-30; higher score indicating more dysfunction). The areas of sexual functioning included were total score used as a global measure of sexual dysfunction. A follow-up version of the questionnaire includes an additional sixth item of the participant's global impression of improvement, with a score ranging from 1 to 6. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: Female participants from all subject population used. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 47 | 52
Score on a scale
  Total score, Week 1: number analyzed (Participants) | 3 | 2
  Total score, Week 1 | -0.3 (0.58) | 0.5 (4.95)
  Total score, Week 2: number analyzed (Participants) | 3 | 5
  Total score, Week 2 | 1.0 (3.61) | 0.2 (4.32)
  Total score, Week 4: number analyzed (Participants) | 34 | 37
  Total score, Week 4 | -1.1 (4.42) | -1.4 (5.23)
  Total score, Week 6: number analyzed (Participants) | 6 | 4
  Total score, Week 6 | -1.3 (7.23) | 0.5 (3.79)
  Total score, Week 8: number analyzed (Participants) | 25 | 18
  Total score, Week 8 | -1.4 (4.90) | -2.1 (4.66)
  Total score, Week 10: number analyzed (Participants) | 5 | 5
  Total score, Week 10 | -1.0 (2.24) | -2.4 (2.61)
  Total score, Week 12: number analyzed (Participants) | 18 | 9
  Total score, Week 12 | -2.9 (5.84) | -1.0 (4.30)

21. Secondary Outcome: Change From Baseline in MSFQ Items (Diminished/Absent Libido; Arousal Difficulties; Orgasm Difficulties/Anorgasmia and Degree of Sexual Satisfaction) Scores
Description: The MSFQ was derived from the Guided Interview Questionnaire for males and from the Arizona Sexual Experience Scale. The questionnaire includes five items with a score ranging from 1-6 (1: greater than normal; 2: normal; 3: minimally diminished; 4: moderately diminished; 5: markedly diminished and 6: totally absent). The areas of sexual functioning included were diminished/absent libido; arousal difficulties; orgasm difficulties/anorgasmia and degree of sexual satisfaction. A follow-up version of the questionnaire includes an additional sixth item of the participant's global impression of improvement, with a score ranging from 1 to 6. It was assessed at Baseline, Week 1, 2, 4, 6, 8, 10 and 12. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as value on Day 1 (pre-dose).
Time Frame: Baseline (Day 1 pre-dose) and up to Week 12
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 60 | 69
Score on a scale
  Absent libido score, Week 1: number analyzed (Participants) | 4 | 2
  Absent libido score, Week 1 | -0.3 (0.50) | 1.0 (1.41)
  Absent libido score, Week 2: number analyzed (Participants) | 6 | 5
  Absent libido score, Week 2 | 0.2 (0.75) | -0.2 (1.48)
  Absent libido score, Week 4: number analyzed (Participants) | 42 | 48
  Absent libido score, Week 4 | -0.3 (1.15) | -0.2 (1.65)
  Absent libido score, Week 6: number analyzed (Participants) | 7 | 7
  Absent libido score, Week 6 | -0.3 (1.98) | 0.6 (1.51)
  Absent libido score, Week 8: number analyzed (Participants) | 30 | 27
  Absent libido score, Week 8 | -0.4 (1.38) | -0.6 (1.28)
  Absent libido score, Week 10: number analyzed (Participants) | 6 | 8
  Absent libido score, Week 10 | 0.2 (0.41) | -0.6 (0.74)
  Absent libido score, Week 12: number analyzed (Participants) | 21 | 15
  Absent libido score, Week 12 | -0.6 (1.77) | -0.4 (1.06)
  Arousal difficulties score, Week 1: number analyzed (Participants) | 4 | 2
  Arousal difficulties score, Week 1 | 0.0 (0.00) | 0.0 (0.00)
  Arousal difficulties score, Week 2: number analyzed (Participants) | 6 | 5
  Arousal difficulties score, Week 2 | 0.3 (0.52) | 0.4 (0.89)
  Arousal difficulties score, Week 4: number analyzed (Participants) | 42 | 48
  Arousal difficulties score, Week 4 | -0.3 (1.18) | -0.3 (1.14)
  Arousal difficulties score, Week 6: number analyzed (Participants) | 7 | 7
  Arousal difficulties score, Week 6 | 0.0 (1.83) | 0.3 (0.49)
  Arousal difficulties score, Week 8: number analyzed (Participants) | 30 | 27
  Arousal difficulties score, Week 8 | -0.4 (1.33) | -0.6 (1.22)
  Arousal difficulties score, Week 10: number analyzed (Participants) | 6 | 8
  Arousal difficulties score, Week 10 | 0.0 (0.00) | -0.8 (1.04)
  Arousal difficulties score, Week 12: number analyzed (Participants) | 21 | 15
  Arousal difficulties score, Week 12 | -0.6 (1.53) | -0.3 (1.39)
  Anorgasmia score, Week 1: number analyzed (Participants) | 4 | 2
  Anorgasmia score, Week 1 | 0.0 (0.00) | -0.5 (2.12)
  Anorgasmia score, Week 2: number analyzed (Participants) | 6 | 5
  Anorgasmia score, Week 2 | -0.7 (2.42) | -0.4 (1.52)
  Anorgasmia score, Week 4: number analyzed (Participants) | 42 | 48
  Anorgasmia score, Week 4 | -0.2 (1.01) | -0.2 (1.38)
  Anorgasmia score, Week 6: number analyzed (Participants) | 7 | 7
  Anorgasmia score, Week 6 | 0.0 (1.53) | 0.3 (1.38)
  Anorgasmia score, Week 8: number analyzed (Participants) | 30 | 27
  Anorgasmia score, Week 8 | -0.2 (1.13) | -0.6 (1.31)
  Anorgasmia score, Week 10: number analyzed (Participants) | 6 | 8
  Anorgasmia score, Week 10 | -0.5 (1.22) | -1.1 (1.36)
  Anorgasmia score, Week 12: number analyzed (Participants) | 21 | 15
  Anorgasmia score, Week 12 | -0.4 (1.63) | -0.4 (1.18)
  Sexual satisfaction score, Week 1: number analyzed (Participants) | 4 | 2
  Sexual satisfaction score, Week 1 | -0.3 (0.50) | 0.0 (1.41)
  Sexual satisfaction score, Week 2: number analyzed (Participants) | 6 | 5
  Sexual satisfaction score, Week 2 | -0.3 (1.51) | 0.4 (0.89)
  Sexual satisfaction score, Week 4: number analyzed (Participants) | 42 | 48
  Sexual satisfaction score, Week 4 | -0.1 (1.22) | -0.5 (1.47)
  Sexual satisfaction score, Week 6: number analyzed (Participants) | 7 | 7
  Sexual satisfaction score, Week 6 | 0.0 (3.00) | -0.3 (0.49)
  Sexual satisfaction score, Week 8: number analyzed (Participants) | 30 | 27
  Sexual satisfaction score, Week 8 | -0.4 (1.10) | -0.6 (1.45)
  Sexual satisfaction score, Week 10: number analyzed (Participants) | 6 | 8
  Sexual satisfaction score, Week 10 | -0.5 (0.84) | -1.3 (1.16)
  Sexual satisfaction score, Week 12: number analyzed (Participants) | 21 | 15
  Sexual satisfaction score, Week 12 | -0.6 (1.63) | -0.5 (1.30)

22. Secondary Outcome: Number of Participant With Suicidal Behavior Based on the Columbia Suicide Severity Rating Scale (C-SSRS) During and Post Treatment
Description: The C-SSRS used to assess severity and change of suicidality by integrating both behavior and ideation and to be completed by the participants. The SSRS track change in the severity/density of suicidality. The interview was initiated with 5 (yes/no) questions; rated on 1-5 point scale, presented in ascending order of severity, about suicidal ideation. If the answers to the first 2 ideation questions were "yes," the clinician asked questions 3-5. If the answers to ideation questions 1 and 2 were "no," then the clinician proceeded to 5 (yes/no) questions that addressed suicidal behavior, which was categorized as actual attempt, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt and preparatory acts or behaviors. Participants analyzed were number of participants with at least one C-SSRS assessment after the first dose of study medication (that is on treatment or post treatment).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12 and Day 14 of follow-up (approximately 14 weeks)
Population: All subject population. Only those participants available at the time of indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 59 | 68
Participants
  Actual attempt | 1 | 1
  Engaged in non-suicidal self-injurious behavior | 1 | 1
  Interrupted attempt | 2 | 1
  Aborted attempt | 1 | 1
  Preparatory acts or behaviors | 0 | 1

23. Secondary Outcome: Number of Participant by Maximum Suicidal Ideation, Based on the C-SSRS During and Post Treatment
Description: The C-SSRS used to assess severity and change of suicidality by integrating both behavior and ideation and to be completed by the participants. The SSRS track change in the severity/density of suicidality. It assessed intensity of ideation (a potentially important marker of severity), specifically asking about frequency, duration, intrusiveness, controllability, and deterrents. The interview was initiated with 5 (yes/no) questions; rated on 1-5 point scale, presented in ascending order of severity, about suicidal ideation. The clinician asked 5 questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation without intent to act, active suicidal ideation with any methods (not plan) without intent to act and active suicidal ideation with specific plan and intent. Participants analyzed were number of participants with at least one C-SSRS assessment after the first dose of study medication (that is on treatment or post treatment).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12 and Day 14 of follow-up (approximately 14 weeks)
Population: All subject population. Only those participants available at the time of indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
Number analyzed (Participants) | 59 | 68
Participants
  Wish to be dead | 9 | 9
  Non-specific active suicidal thoughts | 2 | 4
  Active suicidal ideation without intent to act | 1 | 0
  Active suicidal ideation with any methods | 1 | 0
  Active suicidal ideation with plan and intent | 1 | 0

ADVERSE EVENTS:
Time Frame: AE and SAE were reported from the start of investigational product and until the follow-up contact (up to 18 weeks).
Description: All subject population was used for the analysis of safety (AE and SAE).
Arm/Group | Placebo | Orvepitant 60 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/69
Other Adverse Events (participants affected / at risk) | 27/60 | 34/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Orvepitant 60 mg Once Daily (N=69)
Convulsion (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Orvepitant 60 mg Once Daily (N=69)
Headache (Nervous system disorders) | 8 (8) | 11 (13)
Nausea (Gastrointestinal disorders) | 6 (7) | 7 (8)
Somnolence (Nervous system disorders) | 3 (3) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (3)
Fatigue (General disorders) | 3 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated on 11 May 2010 upon the recommendation of the Data Safety Monitoring Board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.